CLINICAL TRIAL: NCT06430775
Title: Exploring Prolonged Arthrogenic Muscle Responses and Associated Factors After Anterior Cruciate Ligament Reconstruction
Brief Title: Exploring Prolonged AMR in ACL Reconstructed Patients
Status: Recruiting | Type: Observational
Sponsor: University Ghent (Other)
Collaborators: Research Foundation Flanders (Other)
Responsible Party: Sponsor
Other Study IDs: G086223N; ONZ-2023-0365 (Other: Ethical committee Ghent University)
Record Dates: First submitted 2024-05-17; First posted 2024-05-28 (Actual); Last update posted 2024-07-01 (Actual); Status verified 2024-06

CONDITIONS: Anterior Cruciate Ligament Injuries; Anterior Cruciate Ligament Rupture; Anterior Cruciate Ligament Tear; ACL; ACL Injury; ACL Tear; Anterior Cruciate Ligament Reconstruction; Arthrogenic Muscle Inhibition; Arthrogenic Muscle Responses
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- ACLR-patients: The participants to be studied will have an anterior cruciate ligament injury for which surgical treatment is scheduled.

SUMMARY:
The goal of this observational study is to explore the significance of subject-reported outcomes and clinical parameters in relation to the occurence of prolonged presence of arthrogenic muscle responses (AMR) in anterior cruciate ligament (ACL) reconstructed patients. The main questions it aims to answer are:

1. Is there a link between the long-term occurence of AMR in ACL reconstructed patients and the level of kinesiophobia experienced before or after their ACL surgery? We hypothesize that ACL patients with higher levels of kinesiophobia are more likely to exhibit prolonged AMR as an unconscious reaction to protect their affected knee joint.

2. Is the long-term presence of AMR in ACL reconstructed patients linked to their subjective knee function and stability (at certain time points throughout their recovery)? Our hypothesis is that poorer subjective knee function and stability might be associated with the presence of prolonged arthrogenic muscle responses in ACL reconstructed patients.

3. Is the prolonged presence of AMR in ACL reconstructed patients linked to their pain levels (at certain time points throughout their recovery)? Our hypothesis is that ACL patients with higher pre- and/or postsurgical pain levels may exhibit a higher degree of long-lasting AMR.

4. Is the long-term presence of AMR in ACL reconstructed patients linked to clinical parameters such as swelling, isometric quadriceps and hamstrings strength and knee range of motion (at certain time points throughout their recovery)? Our hypothesis is that ACL patients with poorer outcomes in terms of these clinical parameters may be more likely to exhibit prolonged AMR.

Participants will:

* Fill in the following questionnaires 1 week before surgery and at 1 and 3 months after surgery:

  * Demopgraphical information
  * Knee Injury and Osteoarthritis Outcome Score (KOOS)
  * Lysholm Score (only question 1)
  * Tegner Activity Scale (current activity level, pre-injury activity level and desired activity level after recovery)
  * Numeric Rating Score (NRS) for pain levels during the day & during the night
  * ACL-Return to Sport after Injury Scale (ACL-RSI)
* Complete a testing protocol 5 months after their surgery, which includes bilateral electromyographical measurements of the hamstrings and quadriceps during jumping tasks and a quadriceps inhibition measurement using the interpolated twitch method to evaluate the presence of prolonged AMR.

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years old.
* Having suffered an ACL rupture.
* Undergoing a surgical ACL reconstruction in the AZ Delta hospital in Roeselare (Campus Brugsesteenweg).

Exclusion Criteria:

* Revision ACL reconstruction.
* Other severe injuries to the lower limbs within the past year.
* Muscular or neurological disorders affecting lower limb functioning.
* Fibromyalgia or chronic fatigue syndrome.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients aged between 18 and 40 who have suffered an ACL rupture and for whom ACL reconstructive surgery is planned at AZ Delta Hospital in Roeselare.
Sampling Method: Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2023-10-15 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Voluntary quadriceps activation | 5 months post ACL reconstruction
  A torque-based isometric biodex measurement using the interpolated twitch technique.
Quadriceps and hamstrings activity / cocontraction during jumping tasks | 5 months post ACL reconstruction
  Electromyographical measurement of quadriceps and hamstrings activation during jumping tasks: bilateral countermovement jump, unilateral countermovement jump and unilateral vertical drop jump with a 90° medial turn. The cocontraction will be quantified with cocontraction indices.

SECONDARY OUTCOMES:
Quadriceps strength | 5 months post ACL reconstruction
  Concentric and isokinetic Biodex measurements of the quadriceps strength
Hamstrings strength | 5 months post ACL reconstruction
  Concentric and isokinetic Biodex measurements of the quadriceps strength
Patient reported knee function | 5 months post ACL reconstruction
  Questioned using the Knee Injury and Osteoarthritis Outcome Score (KOOS). Scores on the KOOS range from 0-100, with 0 representing the greatest possible problems in terms of knee function and 100 representing no problems.

CONTACTS AND LOCATIONS:
Locations (1):
- AZ Delta Hospital (Campus Brugsesteenweg), Roeselare, West-Vlaanderen, Belgium

IPD SHARING:
Plan to Share IPD: Yes
All collected IPD that underlie results in a publication will be shared.
Supporting Information: Study Protocol, SAP
Time Frame: The data will become available after publication.